CLINICAL TRIAL: NCT02589197
Title: Muscle Activation and Biomechanical Function of the Lower-limb Joints Following Total Knee Arthroplasty With Medial-pivot or Posterior-stabilized Implants: an Electromyography Study
Brief Title: Gait and Functional Outcomes Study Following Total Knee Arthroplasty With Medial-pivot or Posterior-stabilized Implants
Acronym: GOLD
Status: Completed | Type: Observational
Sponsor: MicroPort Orthopedics Inc. (Industry)
Collaborators: University of Ottawa (Other); The Ottawa Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 15-LJK-001
Record Dates: First submitted 2015-10-19; First posted 2015-10-28 (Estimated); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Joint Disease
Keywords: osteoarthritis; correction of functional deformity; procedures; traumatic osteoarthritis; degenerative osteoarthritis; total knee arthroplasty; Healthy Volunteers; electromyography; Musculoskeletal Diseases
MeSH Terms: conditions — Joint Diseases; Osteoarthritis; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1 (Medial-Pivot): Group 1 will be implanted with the EVOLUTION® MP System with Cruciate Sacrificing (CS) tibial inserts.
  Interventions: Device: Group 1 (Medial-Pivot)
- Group 2 (Posterior-Stabilized): Group 2 will be implanted with the Zimmer® NexGen® PS TKA system.
  Interventions: Device: Group 2 (Posterior-Stabilized)
- Group 3 (Control Group): Non-implanted control subjects

INTERVENTIONS:
Device: Group 1 (Medial-Pivot) — EVOLUTION® Total Knee Arthroplasty Medial Pivot system with CS inserts
  Other Names: EVOLUTION® CS TKA System; Total Knee Arthroplasty Sytem; EVOLUTION®
  Groups: Group 1 (Medial-Pivot)
Device: Group 2 (Posterior-Stabilized) — Zimmer® NexGen® Total Knee Arthroplasty system with PS inserts
  Other Names: Zimmer® NexGen® PS TKA System; Total Knee Arthroplasty Sytem; NexGen®
  Groups: Group 2 (Posterior-Stabilized)

SUMMARY:
MicroPort Orthopedics (MPO) is conducting this study to build upon the results of a previous study which showed the Medial Pivot (MP) system required lower quadriceps activation than subjects implanted with a Posterior stabilized (PS) system preforming the same activities of daily living.

DETAILED DESCRIPTION:
MicroPort Orthopedics (MPO) is conducting this study to build upon the results of a previous study which showed the Medial Pivot (MP) system required lower quadriceps activation than subjects implanted with a Posterior stabilized (PS) system preforming the same activities of daily living. The propose of the current study is to determine the impact of Total Knee Arthroplasty (TKA) design on muscle activation following TKA surgery.

ELIGIBILITY:
Inclusion Criteria:

To be included in Groups 1 and 2, subjects must meet all of the following criteria:

Subject is a candidate for unilateral primary TKA for degenerative or traumatic osteoarthritis Subject is a candidate to be implanted with the specified combination of components for either Group 1 or 2 Subjects are at least 45 years old and less than 76 years of age at time of enrollment Subject is willing and able to complete required study visits and assessments Subject plans to be available through the 1 year postoperative follow-up visit Subject is willing to sign the approved Informed Consent document

To be included in Group 3, subjects must meet all of the following criteria:

Subjects are at least 45 years old and less than 76 years of age at time of enrollment Subject is willing and able to complete required study visit and assessments Subject is willing to sign the approved Informed Consent document

Exclusion Criteria:

Subjects will be excluded if they meet any of the following criteria:

Subject has both a body mass index (BMI) and waist circumference measurements greater than 35.0 kg/m2 and 102.0 cm respectively for men and 35.0 kg/m2 and 88.0 cm respectively for women at screening.

Groups 1 & 2 Only: Subject has degenerative conditions (other than osteoarthritis in the enrolled TKA) impacting joints of the lower extremities, previous joint replacement of the enrolled knee or other lower limb joint replacement, or any other past or present condition, which in the opinion of the Investigator may impact gait. Group 3 Only: Subject has degenerative condition impacting joints of the lower extremities, any previous joint replacement in the knees, or any other past or present condition, which in the opinion of the Investigator may impact gait.

Groups 1 and 2 Only: Subjects with a Kellgren-Lawrence Grading Scale of ≥2 on the contralateral knee if having severe pain or abnormal gait patterns.

Subject is currently enrolled in another clinical investigation related to lower limbs which could affect the endpoints of this protocol.

Subject is unwilling or unable to sign the Informed Consent document Subject has documented substance abuse issues Subject has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study Subject is currently incarcerated or has impending incarceration

Ages: 45 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will be selected from the orthopedic clinic at The Ottawa hospital for implanted patients. Non-implanted subjects will be selected from the community.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-07-13 (Actual); Primary Completion 2022-09 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Lower Limb Muscle Activation Comparison as Assessed by Maximum Voluntary Isometric Contraction Muscle Strength and Dynamic Muscle Activation Measurements in Total Knee Arthroplasty Subjects Implanted with Medial-pivot or Posterior-stabilized Implants | Presurgery and 12 Months Post Surgery
  Measured by Dynamic Muscle Activation Measurements and Maximum Voluntary Isometric Contraction Muscle Strength and Activation

SECONDARY OUTCOMES:
Compare lower limb muscle activation between the control group (Group 3) and Groups 1 and 2, as assessed by maximum voluntary isometric contraction muscled strength and dynamic muscle activation measurements | Presurgery and 12 Months Post Surgery for implanted subjects
  Measured by Dynamic Muscle Activation Measurements and Maximum Voluntary Isometric Contraction Muscle Strength and Activation
Compare functional outcomes for the Groups 1 and 2 as assessed by the Timed Up & Go (TUG) test | Presurgery and 12 Months Post Surgery for implanted subjects
  Measured by Timed Up & Go (TUG) test
Compare functional outcomes for the Groups 1 and 2 as assessed by the KOOS Scores | Presurgery and 12 Months Post Surgery for implanted subjects
  Measured by KOOS Scores
Compare subject satisfaction using a custom five question patient satisfaction questionnaire for Groups 1 and 2 | 12 Months Post Surgery
  Measured by Patient Satisfaction Survey

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Dervin, MD, Principal Investigator — Ottawa Hospital
Locations (2):
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - University of Ottawa, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kowalski E, Catelli DS, Pelegrinelli ARM, Dervin G, Lamontagne M. EFORT Michael Freeman Award 2020: Knee biomechanics before and after total knee arthroplasty with either a medial pivot or posterior stabilized implants. Clin Biomech (Bristol). 2025 Jul;127:106604. doi: 10.1016/j.clinbiomech.2025.106604. Epub 2025 Jun 26. PMID 40602029